CLINICAL TRIAL: NCT00424294
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Of CP-195543 And Celecoxib Dual Therapy In The Treatment Of The Signs And Symptoms Of Rheumatoid Arthritis In Subjects Who Are Inadequately Controlled On Methotrexate
Brief Title: A Study Of CP-195543 And Celecoxib Dual Therapy In Subjects With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See Detailed Description field
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A7701005
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Celecoxib; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Celecoxib (Active Comparator): Celecoxib with placebo therapy.
  Interventions: Drug: celecoxib
- Methotrexate (Other): Background Methotrexate taken in both CP-195,543/Celecoxib and Celecoxib only arms.
  Interventions: Drug: Methotrexate
- CP-195,543 (Experimental): CP-195,543 and Celecoxib dual therapy.
  Interventions: Drug: CP-195,543

INTERVENTIONS:
Drug: CP-195,543 — CP-195543 is a potent and specific antagonist of the leukotriene B4 (LTB4) receptor.
  Arms: CP-195,543
Drug: celecoxib — Celecoxib is a nonsteroidal anit-inflammatory drug (NSAID) marketed worldwide (in the United States [US] as Celeberex) and approved for the relief of signs and symptoms of osteoarthritis.
  Arms: Celecoxib
Drug: Methotrexate — Methotrexate is a folate analogue that, based on it efficacy and safety in RA, is commonly used as frontline DMARD treatment in patients with moderate to severe disease who do not respond to NSAIDs alone.
  Arms: Methotrexate

SUMMARY:
To evaluate the efficacy, safety and tolerability of CP-195543 and celecoxib dual therapy in subjects with rheumatoid arthritis

DETAILED DESCRIPTION:
Trial enrollment was prematurely discontinued on December 3, 2007. The results of an interim efficacy and safety analysis demonstrated an overall poor tolerability profile and high discontinuation rate when dual therapy with CP-195543 and Celecoxib was administered. The decision to discontinue further enrollment in the trial was not based on any efficacy or serious safety concerns. Previously enrolled study participants continued in the study and the trial completed on February 27, 2008.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of RA based upon the American college of Rheumatology 1987 revised criteria
* Active disease at Screening
* Stable dose of methotrexate between 10-25 mg/week oral or parenteral

Exclusion Criteria:

* A diagnosis of any other inflammatory or secondary, noninflammatory arthritis that, in the opinion of the Investigator, would interfere with disease activity assessments
* A history of hypersensitivity or allergic type reactions to cyclooxygenase inhibitors, opiates, aspirin or sulfonamides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (38):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Dunedin, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Lake Mary, Florida
  - Pfizer Investigational Site, Miramar, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Orange City, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Port Richey, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Venice, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, Moline, Illinois
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Munster, Indiana
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Covington, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Frederick, Maryland
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Olean, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Philladelphia, Pennsylvania
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Killeen, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Ogden, Utah

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7701005&StudyName=A%20Study%20Of%20CP-195543%20And%20Celecoxib%20Dual%20Therapy%20In%20Subjects%20With%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo and Celecoxib: Placebo matched to CP-195543 capsule orally twice daily along with celecoxib capsule 200 milligram (mg) orally twice daily for 12 weeks. A stable dose of methotrexate greater than or equal to (>=) 10 milligram per week (mg/week) and less than or equal to (<=) 25 mg/week via oral or parenteral route was continued as background therapy.
- CP-195543 and Celecoxib: CP-195543 capsule 400 mg orally twice daily along with celecoxib capsule 200 mg orally twice daily for 12 weeks. A stable dose of methotrexate >=10 mg/week and <=25 mg/week via oral or parenteral route was continued as background therapy.
Period: Overall Study
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Started | 36 | 34
Treated | 35 | 34
Completed | 28 | 19
Not Completed | 8 | 15
Not completed — Adverse Event | 4 | 10
Not completed — Lack of Efficacy | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Other | 0 | 2
Not completed — Randomized but not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) was an intent-to-treat analysis set including all participants randomized to treatment who had taken at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (11.6) | 57.7 (12.7) | 55.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 27 | 60
  Male | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 12
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in tender joint count; >=20% improvement in swollen joint count; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 12
Population: FAS was an intent-to-treat analysis set including all participants randomized to treatment who had taken at least 1 dose of study drug. Missing values were imputed using last observation carried forward (LOCF) method.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
percentage of participants | 31.43 | 35.29
Statistical Analysis 1: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Test type: Superiority or Other; p = 0.733, Chi-squared

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 1, 2, 4 and 8
Description: ACR20 response: >=20% improvement in tender joint count; >=20% improvement in swollen joint count; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 1, 2, 4, 8
Population: FAS was an intent-to-treat analysis set including all participants randomized to treatment who had taken at least 1 dose of study drug. Missing values were imputed using LOCF method.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
percentage of participants
  Week 1 | 31.43 | 23.53
  Week 2 | 28.57 | 35.29
  Week 4 | 28.57 | 41.18
  Week 8 | 25.71 | 38.24
Statistical Analysis 1: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 1: p-value was calculated by Chi-square test; Test type: Superiority or Other; p = 0.463, Chi-squared
Statistical Analysis 2: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 2: p-value was calculated by Chi-square test; Test type: Superiority or Other; p = 0.549, Chi-squared
Statistical Analysis 3: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 4: p-value was calculated by Chi-square test; Test type: Superiority or Other; p = 0.272, Chi-squared
Statistical Analysis 4: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 8: p-value was calculated by Chi-square test; Test type: Superiority or Other; p = 0.265, Chi-squared

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: >=50% improvement in tender joint count; >=50% improvement in swollen joint count; and >=50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 1, 2, 4, 8, 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
percentage of participants
  Week 1 | 0.0 | 0.0
  Week 2 | 0.0 | 0.0
  Week 4 | 8.57 | 2.94
  Week 8 | 5.71 | 11.76
  Week 12 | 8.57 | 14.71
Statistical Analysis 1: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 4: p-value was calculated by Fisher exact test; Test type: Superiority or Other; p = 0.939, Fisher Exact
Statistical Analysis 2: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 8: p-value was calculated by Fisher exact test; Test type: Superiority or Other; p = 0.323, Fisher Exact
Statistical Analysis 3: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 12: p-value was calculated by Fisher exact test; Test type: Superiority or Other; p = 0.338, Fisher Exact

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: >=70% improvement in tender joint count; >=70% improvement in swollen joint count; and >=70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 1, 2, 4, 8, 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
percentage of participants
  Week 1 | 0.0 | 0.0
  Week 2 | 0.0 | 0.0
  Week 4 | 0.0 | 0.0
  Week 8 | 0.0 | 0.0
  Week 12 | 2.86 | 2.94
Statistical Analysis 1: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 12: p-value was calculated by Fisher exact test; Test type: Superiority or Other; p = 0.746, Fisher Exact

5. Secondary Outcome: Change From Baseline in Tender/Painful Joint Count (TJC) at Week 1, 2, 4, 8 and 12
Description: Participants were assessed for tender/painful joints using a 28-joint count comprised of left and right shoulders, elbows, wrists, proximal interphalangeal joints, metacarpophalangeal joints and knees. Artificial joints were not assessed.
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: FAS was an intent-to-treat analysis set including all participants randomized to treatment who had taken at least 1 dose of study drug.Here,"n" signifies those participants who were evaluable at specified time point for each arm,respectively. For descriptive data,observed cases were reported and for statistical data,LOCF imputation method was used.
Measure: Mean (Standard Deviation); unit: tender/painful joints
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
tender/painful joints
  Baseline (n=35, 34) | 15.54 (5.55) | 13.74 (7.15)
  Change at Week 1 (n=33, 31) | -4.45 (5.15) | -4.68 (6.29)
  Change at Week 2 (n=34, 31) | -3.82 (6.24) | -6.13 (6.15)
  Change at Week 4 (n=31, 25) | -5.68 (6.48) | -5.04 (6.09)
  Change at Week 8 (n=33, 24) | -5.15 (6.46) | -6.00 (7.68)
  Change at Week 12 (n=30, 21) | -5.67 (5.86) | -5.95 (9.45)
Statistical Analysis 1: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 1: Analysis of covariance (ANCOVA) with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.635, ANCOVA
Statistical Analysis 2: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 2: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.044, ANCOVA
Statistical Analysis 3: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 4: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.957, ANCOVA
Statistical Analysis 4: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 8: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.597, ANCOVA
Statistical Analysis 5: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 12: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.960, ANCOVA

6. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) at Week 1, 2, 4, 8 and 12
Description: Participants were assessed for swollen joints using a 28-joint count comprised of left and right shoulders, elbows, wrists, proximal interphalangeal joints, metacarpophalangeal joints and knees. Artificial joints were not assessed.
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
swollen joints
  Baseline (n=35, 34) | 11.49 (4.85) | 12.00 (5.75)
  Change at Week 1 (n=33, 31) | -3.18 (4.23) | -4.35 (4.41)
  Change at Week 2 (n=34, 31) | -2.74 (5.59) | -5.97 (5.27)
  Change at Week 4 (n=31, 25) | -3.45 (6.20) | -6.32 (4.71)
  Change at Week 8 (n=33, 24) | -2.79 (6.38) | -6.71 (5.44)
  Change at Week 12 (n=30, 21) | -3.80 (6.70) | -6.38 (6.10)
Statistical Analysis 1: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 1: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.252, ANCOVA
Statistical Analysis 2: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 2: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.032, ANCOVA
Statistical Analysis 3: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 4: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.031, ANCOVA
Statistical Analysis 4: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 8: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.018, ANCOVA
Statistical Analysis 5: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.170, ANCOVA

7. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain at Week 1, 2, 4, 8 and 12
Description: Patient's assessment of arthritis pain was assessed using a 100 millimeter (mm) visual analogue scale (VAS) with range: 0 = no pain to 100 = worst possible pain.
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
mm
  Baseline (n=35, 34) | 50.94 (23.36) | 54.74 (22.25)
  Change at Week 1 (n=33, 30) | -13.27 (20.21) | -11.33 (15.97)
  Change at Week 2 (n=34, 32) | -9.53 (23.98) | -9.50 (23.65)
  Change at Week 4 (n=31, 25) | -8.16 (23.62) | -14.12 (24.97)
  Change at Week 8 (n=33, 24) | -14.06 (24.82) | -12.04 (29.37)
  Change at Week 12 (n=30, 21) | -11.50 (22.90) | -21.43 (35.24)
Statistical Analysis 1: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 1: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.507, ANCOVA
Statistical Analysis 2: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 2: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.743, ANCOVA
Statistical Analysis 3: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 4: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.914, ANCOVA
Statistical Analysis 4: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 8: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.715, ANCOVA
Statistical Analysis 5: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.558, ANCOVA

8. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Arthritis at Week 1, 2, 4, 8 and 12
Description: Patient's global assessment of arthritic condition assessed all the ways participants' illness and health conditions affect them at the time of assessment. The response was scored on a 5-point scale: 1 = Very Good (Asymptomatic and no limitation of normal activities), 2 = Good (Mild symptoms and no limitation of normal activities), 3 = Fair (Moderate symptoms and limitation of some normal activities), 4 = Poor (Severe symptoms and inability to carry out most normal activities) and 5 = Very Poor (Very severe symptoms which are intolerable and inability to carry out all normal activities).
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
units on a scale
  Baseline (n=35, 34) | 3.14 (0.88) | 3.24 (0.89)
  Change at Week 1 (n=33, 31) | -0.58 (0.83) | -0.48 (0.89)
  Change at Week 2 (n=34, 31) | -0.38 (0.92) | -0.61 (0.95)
  Change at Week 4 (n=31, 25) | -0.39 (0.95) | -0.68 (0.95)
  Change at Week 8 (n=33, 24) | -0.58 (0.90) | -0.46 (1.02)
  Change at Week 12 (n=30, 21) | -0.40 (1.22) | -0.57 (1.33)
Statistical Analysis 1: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 1: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.172, ANCOVA
Statistical Analysis 2: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 2: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.738, ANCOVA
Statistical Analysis 3: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 4: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.948, ANCOVA
Statistical Analysis 4: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 8: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.428, ANCOVA
Statistical Analysis 5: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.861, ANCOVA

9. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Arthritis at Week 1, 2, 4, 8 and 12
Description: Investigator assessed overall appearance of arthritis at the time of the visit. The response was scored on a 5-point scale: 1 = Very Good (Asymptomatic and no limitation of normal activities), 2 = Good (Mild symptoms and no limitation of normal activities), 3 = Fair (Moderate symptoms and limitation of some normal activities), 4 = Poor (Severe symptoms and inability to carry out most normal activities) and 5 = Very Poor (Very severe symptoms which are intolerable and inability to carry out all normal activities).
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
units on a scale
  Baseline (n=35, 34) | 3.37 (0.49) | 3.32 (0.59)
  Change at Week 1 (n=33, 31) | -0.76 (0.61) | -0.58 (0.67)
  Change at Week 2 (n=34, 31) | -0.74 (0.83) | -0.58 (0.76)
  Change at Week 4 (n=31, 25) | -0.71 (0.94) | -0.60 (0.71)
  Change at Week 8 (n=33, 24) | -0.67 (1.05) | -0.71 (0.69)
  Change at Week 12 (n=30, 21) | -0.67 (0.99) | -0.67 (1.20)
Statistical Analysis 1: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 1: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.325, ANCOVA
Statistical Analysis 2: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 2: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.386, ANCOVA
Statistical Analysis 3: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 4: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.532, ANCOVA
Statistical Analysis 4: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 8: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.909, ANCOVA
Statistical Analysis 5: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.994, ANCOVA

10. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 1, 2, 4, 8 and 12
Description: Health Assessment Questionnaire-Disability Index (HAQ-DI): participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3, where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
units on a scale
  Baseline (n=34, 34) | 1.65 (0.54) | 1.65 (0.65)
  Change at Week 1 (n=32, 30) | 0.34 (0.43) | -0.18 (0.34)
  Change at Week 2 (n=31, 29) | -0.18 (0.54) | -0.24 (0.38)
  Change at Week 4 (n=30, 25) | -0.34 (0.56) | -0.29 (0.46)
  Change at Week 8 (n=32, 24) | -0.38 (0.67) | -0.30 (0.61)
  Change at Week 12 (n=29, 20) | -0.38 (0.59) | -0.44 (0.78)
Statistical Analysis 1: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 1: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.369, ANCOVA
Statistical Analysis 2: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 2: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.666, ANCOVA
Statistical Analysis 3: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 4: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.530, ANCOVA
Statistical Analysis 4: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 8: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.632, ANCOVA
Statistical Analysis 5: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.801, ANCOVA

11. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Week 1, 2, 4, 8 and 12
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
milligram per deciliter (mg/dL)
  Baseline (n=34, 34) | 0.93 (0.69) | 1.36 (1.35)
  Change at Week 1 (n=32, 31) | -0.06 (0.75) | 0.15 (1.33)
  Change at Week 2 (n=32, 31) | 0.08 (0.66) | 0.61 (2.05)
  Change at Week 4 (n=29, 25) | 0.67 (3.78) | 0.16 (1.35)
  Change at Week 8 (n=32, 24) | 0.15 (0.75) | 0.41 (1.29)
  Change at Week 12 (n=29, 21) | 0.60 (3.47) | 0.03 (0.78)
Statistical Analysis 1: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 1: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.052, ANCOVA
Statistical Analysis 2: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 2: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.108, ANCOVA
Statistical Analysis 3: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 4: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.573, ANCOVA
Statistical Analysis 4: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 8: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.342, ANCOVA
Statistical Analysis 5: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.501, ANCOVA

12. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Week 1, 2, 4, 8 and 12
Description: DAS28-3 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP. It was calculated as DAS28-3 (CRP) = 1.15 + 1.10 * ([0.56 * square root of TJC] + [0.28 * square root of SJC] + [0.36 * natural logarithm of {CRP+1}]). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (CRP) <2.6 = remission.
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
units on a scale
  Baseline (n=34, 34) | 4.78 (0.56) | 4.68 (0.84)
  Change at Week 1 (n=32, 31) | -0.65 (0.66) | -0.71 (0.81)
  Change at Week 2 (n=32, 31) | -0.56 (0.87) | -0.86 (0.72)
  Change at Week 4 (n=29, 25) | -0.82 (1.04) | -0.83 (0.77)
  Change at Week 8 (n=32, 24) | -0.84 (0.96) | -1.04 (1.05)
  Change at Week 12 (n=29, 21) | -0.98 (1.07) | -1.19 (1.40)
Statistical Analysis 1: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 1: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.701, ANCOVA
Statistical Analysis 2: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 2: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.167, ANCOVA
Statistical Analysis 3: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 4: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.948, ANCOVA
Statistical Analysis 4: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 8: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.834, ANCOVA
Statistical Analysis 5: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.977, ANCOVA

13. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Week 1, 2, 4, 8 and 12
Description: Duration of morning stiffness was defined as the time elapsed between the time participant woke up and was able to resume normal activities without stiffness in hours (duration was recorded in hours to the nearest quarter. For those participants with unrelenting stiffness, duration was recorded as 24 hours).
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
hour
  Baseline (n=35, 34) | 2.83 (3.68) | 3.22 (4.34)
  Change at Week 1 (n=33, 31) | -0.11 (1.83) | -0.61 (1.50)
  Change at Week 2 (n=34, 31) | 0.03 (2.16) | -1.34 (4.21)
  Change at Week 4 (n=31, 25) | -0.76 (1.65) | -1.51 (4.53)
  Change at Week 8 (n=33, 24) | 0.34 (4.16) | -1.03 (5.09)
  Change at Week 12 (n=30, 21) | 1.05 (7.61) | -1.65 (5.01)
Statistical Analysis 1: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 1: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.291, ANCOVA
Statistical Analysis 2: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 2: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.080, ANCOVA
Statistical Analysis 3: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 4: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.466, ANCOVA
Statistical Analysis 4: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; Week 8: ANCOVA with treatment and site as independent variables and baseline as the covariate was used for the analysis; Test type: Superiority or Other; p = 0.267, ANCOVA
Statistical Analysis 5: Comparison: Placebo and Celecoxib vs CP-195543 and Celecoxib; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.100, ANCOVA

14. Secondary Outcome: Number of Participants Who Withdrew From Study Due to Lack of Efficacy
Time Frame: Baseline up to Week 12
Population: FAS was an intent-to-treat analysis set including all participants randomized to treatment who had taken at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
participants | 2 | 1

15. Secondary Outcome: Time to Withdrawal Due to Lack of Efficacy
Time Frame: Baseline up to Week 12
Population: Median time and corresponding confidence interval (CI) were not estimable because only less than half of the participants withdrew from study due to lack of efficacy and hence, were insufficient for the analysis.
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 28 days after last dose
Population: Safety analysis set is same as FAS. FAS was an intent-to-treat analysis set including all participants randomized to treatment who had taken at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
participants
  AEs | 29 | 31
  SAEs | 1 | 2

17. Other Pre Specified Outcome: Number of Adverse Events by Severity
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs are classified according to the severity in 3 categories a) mild - AEs does not interfere with participant's usual function b) moderate - AEs interferes to some extent with participant's usual function c) severe - AEs interferes significantly with participant's usual function.
Time Frame: Baseline up to 28 days after last dose
Population: as for outcome 16
Measure: Number; unit: adverse events
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
adverse events
  Mild | 40 | 41
  Moderate | 26 | 25
  Severe | 0 | 5

18. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); liver function (aspartate aminotransferase, alanine aminotransferase, total bilirubin, lactate dehydrogenase, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine, uric acid); electrolytes (sodium, potassium, chloride, calcium, phosphate, bicarbonate); clinical chemistry (glucose, creatine kinase); immunology (CRP); urinalysis (dipstick [urine specific gravity, decimal logarithm of reciprocal of hydrogen ion activity {pH} of urine, glucose, protein, blood, ketones, bilirubin], microscopy [urine RBC, WBC, urate crystals, calcium, oxalate, miscellaneous [urine mucus and leucocytes]).
Time Frame: Baseline up to Week 13
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
participants | 15 | 14

19. Other Pre Specified Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure at Day 7, 14, 21, 28, 42, 56, 84 and 91
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were evaluated in sitting position.
Time Frame: Baseline, Day 7, 14, 21, 28, 42, 56, 84, 91
Population: Safety analysis set is same as FAS. FAS was an intent-to-treat analysis set including all participants randomized to treatment who had taken at least 1 dose of study drug. Here, "n" signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
millimeter of mercury (mmHg)
  Baseline: SBP (n=35, 34) | 123.7 (12.33) | 124.6 (14.97)
  Change at Day 7: SBP (n=33, 30) | -0.2 (12.46) | 0.5 (12.91)
  Change at Day 14: SBP (n=1, 5) | 5.0 (NA) — Standard Deviation (SD) was not calculable as only 1 participant was evaluable at this time point. | 3.2 (4.15)
  Change at Day 21: SBP (n=0, 1) | NA (NA) — Data was not analyzed as there was no participant evaluable for this arm group at the specified time point. | 0.0 (NA) — SD was not calculable as only 1 participant was evaluable at this time point.
  Change at Day 28: SBP (n=1, 2) | 18.0 (NA) — SD was not calculable as only 1 participant was evaluable at this time point. | 0.0 (0.0)
  Change at Day 42: SBP (n=4, 2) | 3.3 (4.57) | 0.0 (28.28)
  Change at Day 56: SBP (n=0, 3) | NA (NA) — Data was not analyzed as there was no participant evaluable for this arm group at the specified time point. | -2.0 (8.00)
  Change at Day 84: SBP (n=27, 17) | 4.7 (13.44) | 6.8 (15.58)
  Change at Day 91: SBP (n=3, 3) | 3.3 (13.65) | -15.7 (12.58)
  Baseline: DBP (n=35, 34) | 77.9 (8.03) | 75.8 (10.81)
  Change at Day 7: DBP (n=33, 30) | -1.3 (8.32) | 1.4 (10.57)
  Change at Day 14: DBP (n=1, 5) | -1.0 (NA) — SD was not calculable as only 1 participant was evaluable at this time point. | 1.2 (7.16)
  Change at Day 21: DBP (n=0, 1) | NA (NA) — Data was not analyzed as there was no participant evaluable for this arm group at the specified time point. | 16.0 (NA) — SD was not calculable as only 1 participant was evaluable at this time point.
  Change at Day 28: DBP (n=1, 2) | -4.0 (NA) — SD was not calculable as only 1 participant was evaluable at this time point. | 8.0 (16.97)
  Change at Day 42: DBP (n=4, 2) | -1.8 (7.76) | -2.0 (11.31)
  Change at Day 56: DBP (n=0, 3) | NA (NA) — Data was not analyzed as there was no participant evaluable for this arm group at the specified time point. | -4.0 (7.21)
  Change at Day 84: DBP (n=27, 17) | 1.4 (7.77) | -0.5 (12.21)
  Change at Day 91: DBP (n=3, 3) | 2.7 (6.43) | -5.3 (4.62)

20. Other Pre Specified Outcome: Change From Baseline in Heart Rate Day 7, 14, 21, 28, 42, 56, 84 and 91
Time Frame: Baseline, Day 7, 14, 21, 28, 42, 56, 84, 91
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
beats per minute
  Baseline (n=35, 34) | 74.3 (7.62) | 74.5 (10.62)
  Change at Day 7 (n=33, 30) | -1.0 (10.00) | 2.2 (9.70)
  Change at Day 14 (n=5, 1) | -3.0 (NA) — SD was not calculable as only 1 participant was evaluable at this time point. | -6.4 (2.19)
  Change at Day 21 (n=0, 1) | NA (NA) — Data was not analyzed as there was no participant evaluable for this arm group at the specified time point. | 2.0 (NA) — SD was not calculable as only 1 participant was evaluable at this time point.
  Change at Day 28 (n=1, 2) | -2.0 (NA) — SD was not calculable as only 1 participant was evaluable at this time point. | 2.0 (8.49)
  Change at Day 42 (n=4, 2) | 3.3 (7.37) | -3.0 (4.24)
  Change at Day 56 (n=0, 3) | NA (NA) — Data was not analyzed as there was no participant evaluable for this arm group at the specified time point. | 7.7 (3.21)
  Change at Day 84 (n=27, 17) | 0.8 (9.41) | 5.1 (14.19)
  Change at Day 91 (n=3, 3) | 1.0 (9.54) | -2.0 (7.21)

21. Other Pre Specified Outcome: Number of Participants With Abnormal Electrocardiogram (ECG)
Description: Criteria for potential clinical concern in ECG parameters: Maximum corrected QT interval (QTc) in range of 450 to less than 480 millisecond (msec), Maximum QTcB interval (Bazett's Correction) (msec) in range of 450 to less than 480 msec, Maximum QTcF interval (Fridericia's Correction) in range of 450 to less than 480 msec, maximum QTc interval increase from baseline in range of 30 to less than 60 msec and >=60 msec.
Time Frame: Baseline up to Week 12
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 34 | 35
participants
  Maximum QTc Interval (msec) | 0 | 7
  Maximum QTcB Interval (Bazett's Correction) | 3 | 9
  Maximum QTcF Interval (Fridericia's Correction) | 0 | 2
  QTcF interval 30 to <60 msec Increase | 1 | 2
  QTcF interval >=60 msec Increase | 0 | 0

22. Other Pre Specified Outcome: Number of Participants With Categorical Vital Signs Data
Description: Number of participants with maximum increase from Baseline in sitting SBP and DBP of greater than or equal to 30 mmHg at Week 12 was reported.
Time Frame: Baseline, Week 12
Population: Safety analysis set is same as FAS. FAS was an intent-to-treat analysis set including all participants randomized to treatment who had taken at least 1 dose of study drug. Detailed categorical data was not estimated since summarized continuous data of the vital signs were considered sufficient for the analysis as per investigator's discretion.
Measure: Number; unit: participants
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Number analyzed (Participants) | 35 | 34
participants
  SBP: >=30 mmHg Increase | 1 | 1
  DBP: >=30 mmHg Increase | 1 | 3

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study. All causality treatment-emergent SAEs and Other AEs were reported.
Arm/Group | Placebo and Celecoxib | CP-195543 and Celecoxib
Serious Adverse Events (participants affected / at risk) | 1/35 | 2/34
Other Adverse Events (participants affected / at risk) | 29/35 | 31/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo and Celecoxib (N=35) | CP-195543 and Celecoxib (N=34)
Coronary artery disease (Cardiac disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo and Celecoxib (N=35) | CP-195543 and Celecoxib (N=34)
Eyelid oedema (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 17
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 4
Haematochezia (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 4
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Chills (General disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Candidiasis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 0
Otitis media (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 6 | 3
Paraesthesia (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early because it was determined that the dual therapy with CP-195543 and celecoxib had poor tolerability and a high discontinuation rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.